CLINICAL TRIAL: NCT01985516
Title: Pain Level During Female Urethral Catheterization - Should we Instill the Lubrication Gel Into the Urethra or Just Lubricate the Catheter's Tip? a Prospective Randomized Study
Brief Title: Female Urethral Catheterization - Instillation of the Lubricating Gel Into the Urethra or Pouring it on the Catheter's Tip?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Assaf Harofeh MC, Dr Kobi Stav, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 132/13
Record Dates: First submitted 2013-10-20; First posted 2013-11-15 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Pain
Keywords: Pain; Urethra; Catheter
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Instillation into the urethra (Experimental): 5mL of 2% lidocaine gel will be instilled directly into the urethra 5 minutes before catheterization
  Interventions: Other: Instillation into the urethra
- Pouring the gel on the tip of the catheter (Active Comparator): 5mL of 2% lidocaine gel will be poured on the distal part of the catheter (from the distal tip to 10 cm proximally)
  Interventions: Other: pouring the gel on the catheter's tip

INTERVENTIONS:
Other: Instillation into the urethra — 5mL of 2% lidocaine gel will be instilled directly into the urethra 5 minutes before catheterization
  Arms: Instillation into the urethra
Other: pouring the gel on the catheter's tip — 5mL of 2% lidocaine gel will be poured on the distal part of the catheter (from the distal tip to 10 cm proximally).
  Arms: Pouring the gel on the tip of the catheter

SUMMARY:
Currently, there are no specific guidelines or best practice suggestions for female catheterization. However, there is a consensus that an anesthetic lubricating gel should be routinely used in women as well.

Urethral lubrication can be performed in two different techniques: instillation of the gel directly into the urethra or pouring the gel on the catheter's tip. In this study, we will evaluate the pain level during female urethral catheterization in each technique.

Our hypothesis is that the level of pain will be much less if the lubrication agent will be instilled directely to the urethra.

DETAILED DESCRIPTION:
This is a randomized prospective study that will compare the pain levels of urethral catheterization in women randomized to intraurethral lidocaine gel instillation or lubrication of the catheter's tip with lidocaine gel.

Women aged 18 years and older who will be referred for multichannel Urodynamic study in order to evaluate lower urinary tract symptomswill be included.

Patients will be randomized to 2 groups: (1) 5mL of 2% lidocaine gel instilled directly into the urethra 5 minutes before catheterization; (2), 5mL of 2% lidocaine gel poured on the distal part of the catheter. The randomization technique will be employed by a computerized random number generator.

A 12F Nelaton urethral catheter will be introduced in order to measure post-void residual volumes. Subsequently, multichannel Urodynamic testing (Duet Encompass System - Mediwatch Group Plc) will be performed using a dual lumen 6F urethral and 9F rectal catheters. Filling will be carried out using room temperature saline at a filling rate of 50 ml/min.

Patients will be requested to fill out a 0 (no pain) to 10 (worst imaginable pain) visual analog pain scale (VAS) in different time points: prior to gel instillation (baseline), immediately after gel instillation (only in group 1), immediately after the introduction of the Nelaton catheter, 5 and 30 minutes after the catheter will be taken out.

Time frame of the study: 30 minutes before the test and 1 hour after the test. Since the study evaluates pain during the procedure the time frame of the study and assessment is very short. longer follow-up is not needed.

ELIGIBILITY:
Inclusion Criteria:

women aged 18 years and older who will be referred for multichannel Urodynamic study in order to evaluate lower urinary tract symptoms.

-

Exclusion Criteria:

use of any analgesics within the previous 24 hours, known urethral stricture, active urinary tract infection, indwelling urethral catheter, pre-existing urethral pain (e.g. patients with chronic pelvic pain syndromes and interstitial cystitis), known allergy to lidocaine or inability to cooperate with pain assessment due to mental disorders.

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in visual analog pain scales | Before instillation, During Instillation of the lubricants, After Urethral Catheterization, 5 and 30 minutes after the catheter removal
  A 0 to 10 visual analog pain scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Kobi Stav, MD, Principal Investigator — Assaf Harofe Medical Center
Locations (1):
- Assaf Harofe Medical Center, Beer Yaakov, Zeriffin, Israel